CLINICAL TRIAL: NCT02216994
Title: Efficacy and Accuracy of a New Diagnostic Scoring System to Differentiate Hirschsprung Disease From Hirschsprung Disease Allied Disorders in the Patients With Suspected Intestinal Dysganglinosis: a Prospective Study
Brief Title: A New Scoring System Improves Diagnostic Accuracy of Intestinal Dysganglionosis --a Prospective Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Collaborators: Jiangxi Province Children's Hospital (Other)
Responsible Party: Principal Investigator, Jiexiong Feng, Director of pediatric surgery department, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TJCD-D-13-00074; tj2014701 (Other: Tongji Hospital)
Record Dates: First submitted 2014-08-06; First posted 2014-08-15 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Hirschsprung Disease
Keywords: Intestinal dysganglinosis; Hirschsprung disease; Hirschsprung disease allied disorders; diagnostic scoring system; Prospective study
MeSH Terms: conditions — Hirschsprung Disease | interventions — Lactulose; Conservative Treatment; Mineral Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- surgery treatment (Other): The patients with a predicting score of more than 5 are diagnosed with HD, and are performed surgery to remove the aganglionic bowel. The patients with a score less than 5 are mostly indicative of HAD, and receive conservative treatments that included colonic irrigation, enema, high dose lactulose, and oral paraffin oil for at least 6 months. When there is no clinical improvement, patients are consented for surgical procedures to remove the dysganglionic bowel segments. one stage pull through procedure to remove the dysganglionic bowel segments.
  Interventions: Drug: high dose lactulose; Behavioral: conservative treatment; Drug: paraffin oil

INTERVENTIONS:
Drug: high dose lactulose — The patients with a score less than 5 are mostly indicative of HAD, and receive conservative therapies that included colonic irrigation, enema, high dose lactulose, and oral paraffin oil for at least 6 months. When there is no clinical improvement, patients are consented for surgical procedures to remove the dysganglionic bowel segments.
  Other Names: Duphalac®
Behavioral: conservative treatment — The patients with a score less than 5 are mostly indicative of HAD, and receive conservative therapies that included colonic irrigation, enema, high dose lactulose, and oral paraffin oil for at least 6 months. When there is no clinical improvement, patients are consented for surgical procedures to remove the dysganglionic bowel segments.
  Other Names: colonic irrigation
Drug: paraffin oil — The patients with a score less than 5 are mostly indicative of HAD, and receive conservative therapies that included colonic irrigation, enema, high dose lactulose, and oral paraffin oil for at least 6 months. When there is no clinical improvement, patients are consented for surgical procedures to remove the dysganglionic bowel segments.
  Other Names: Shilayou®

SUMMARY:
1. The investigators previously reported a simple diagnostic scoring system to differentiate Hirschsprung disease (HD) from Hirschsprung disease allied disorders (HAD) in the patients with suspected intestinal dysganglionosis. In the retrospective study, the investigators concluded that the patients with a predicting score of more than 5 are more likely to be diagnosed with HD, whereas a score less than 5 is mostly indicative of HAD.
2. Since it is essential to confirm the accuracy and efficacy of the scoring system in a prospective manner before it is used as a standard procedure, this prospective study is designed and performed.

DETAILED DESCRIPTION:
1. Patients have hard or firm stools for 2 or less per week, and with ages from newborn to 3 years old are recruited in this study.
2. The recruited patients is undergoing preoperative work-up including barium enema (BE), anorectal manometry (ARM) and histochemical acetylcholinesterase (AChE) staining of rectal mucosa. Known risk factors for intestinal dysganglionosis (IDs) are recorded. The predicting score is calculated by summing the scores of the risk factors and 3 preoperative tests.
3. The patients with a predicting score of more than 5 are diagnosed with HD, and are performed surgery to remove the aganglionic bowel.
4. The patients with a score less than 5 are mostly indicative of HAD, and receive conservative therapies that included colonic irrigation, enema, high dose lactulose, and oral paraffin oil for at least 6 months. When there is no clinical improvement, patients are consented for surgical procedures to remove the dysganglionic bowel segments.

ELIGIBILITY:
Inclusion Criteria:

* Hard or firm stools for 2 or less per week
* Age are from newborn to 3 years old

Exclusion Criteria:

* Children>3 years of age
* Patients presented severe inflammation or malnutrition, unconsciousness or perforation of intestine

Ages: 1 Day to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-12 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
the predicting score calculation | 6-12 months
  The recruited patients is undergoing preoperative work-up including barium enema (BE), anorectal manometry (ARM) and histochemical acetylcholinesterase (AChE) staining of rectal mucosa. Known risk factors for IDs are recorded. The predicting score is calculated by summing the scores of the risk factors and 3 preoperative tests.
  The patients with a predicting score of more than 5 are diagnosed with HD, and are performed surgery to remove the aganglionic bowel.
  The patients with a score less than 5 are mostly indicative of HAD, and receive conservative therapies that included colonic irrigation, enema, high dose lactulose, and oral paraffin oil for at least 6 months. When there is no clinical improvement, patients are consented for surgical procedures to remove the dysganglionic bowel segments.

SECONDARY OUTCOMES:
pathological diagnosis | 12-18 months
  The intestinal specimens were reviewed by 3 experienced pathologists all of whom had participated in a consensus meeting on diagnostic criteria of IDs.

CONTACTS AND LOCATIONS:
Overall Officials: Jiexiong Feng, MD, PhD, Principal Investigator — Tongji Medical College,Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China